CLINICAL TRIAL: NCT07162974
Title: Litholytic Therapy for Coral Urate Nephrolithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSUMD Moscow
Record Dates: First submitted 2025-08-19; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis | interventions — Citric Acid; potassium bicarbonate; Sodium Citrate

STUDY DESIGN:
Intervention Model Description: 49 patients with coral urate stones.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Citrate therapy for coralloid nephrolithiasis (Experimental): Patients were treated with the citrate mixture "Blemaren"
  Interventions: Drug: anhydrous citric acid - 1197.0 mg, potassium bicarbonate - 967.5 mg, sodium citrate anhydrous - 835.5 mg

INTERVENTIONS:
Drug: anhydrous citric acid - 1197.0 mg, potassium bicarbonate - 967.5 mg, sodium citrate anhydrous - 835.5 mg — The dosage was selected individually for each patient, the target pH was considered to be 7.2

SUMMARY:
This is a prospective cohort study, patients with coralloid nephrolithiasis. Purpose of the study: to evaluate the efficacy and safety of litholytic therapy of coral-like urate nephrolithiasis with citrate mixtures.

DETAILED DESCRIPTION:
Anthropometric parameters height and weight were recorded in all patients, body mass index was calculated. All patients underwent MSCT of the urinary tract to assess the volume of density and concrements before the start of therapy. Biochemical blood analysis included determination of creatinine level with subsequent calculation of SCF. Urine pH was monitored for 72 hours using an electronic pH meter before therapy and recorded in a diary by patients three times a day, after which the average pH was calculated. Patients who met the inclusion criteria were included in the study after signing informed consent.

ELIGIBILITY:
* Coral-shaped calculus, which fills one or more calyx and pelvis (K2-K4 according to the classification of coral-shaped concretions);
* The urate composition of the kidney stone was confirmed using dual-energy MSCT;
* Unimpaired or restored (by draining the kidney) urine outflow from the kidney;
* Persistently acidic urine pH (pH 5.8 or less);
* Stone density is 550 Hounsfield units or less;
* Informed voluntary consent of the patient to participate in the study;
* Patient's readiness for conservative treatment;
* No contraindications to therapy with citrate mixtures;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the size, volume and density of stones. | 1 month
  Computer tomography is the "gold standard" for diagnosing urolithiasis; it will allow you to identify stones, determine their size, density, structure, location, and assess the condition of the urinary tract.

SECONDARY OUTCOMES:
Kidney function | 1 month
  Glomerular filtration rate (GFR, ml/min/1.73 m2) is a test used to check how well the kidneys are working. Specifically, it estimates how much blood passes through the glomeruli each minute. A GFR of 60 or higher is in the normal range. A GFR below 60 may mean kidney disease. A GFR of 15 or lower may mean kidney failure.
  The measurement of the glomerular filtration rate will be measured according to the results of the blood test
Assessing the composition of stones | 6 months
  Chemical analysis of stones is a spectrometric (infrared spectroscopy) method that determines its exact composition by analyzing how the stone absorbs infrared radiation. Chemical analysis of stones will be performed on those patients who will undergo surgical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow state university of medicine and dentistry named after A.I. Evdokimov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided